CLINICAL TRIAL: NCT01669850
Title: The Safety and Effectiveness of Clipped Technique vs. Hand-Sewn Technique for Anastomosis in Arteriovenous Fistulas
Brief Title: Clipped Versus Handsewn Arteriovenous Fistula Anastomosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: minimal accrual
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Gundersen Lutheran Health System (Other)
Responsible Party: Principal Investigator, Kara Kallies, Advanced Research Associate, on behalf of Clark Davis, MD (PI), Gundersen Lutheran Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-12-07-002
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Arteriovenous Fistula Complications and Failure
Keywords: Chronic kidney disease; Arteriovenous fistula; Surgical anastomosis; Complications; Patency; Dialysis access
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clipped anastomosis (Experimental): A vascular clip device will be used to create the anastomosis during arteriovenous fistula creation.
  Interventions: Device: Clipped anastomosis
- Handsewn anastomosis (Active Comparator): A handsewn technique will be used to create the anastomosis in arteriovenous fistula creation.
  Interventions: Procedure: Handsewn anastomosis

INTERVENTIONS:
Device: Clipped anastomosis — The vascular clip devise will be used to complete the anastomosis during fistula creation.
  Other Names: Anastoclip (Le Maitre)
  Arms: Clipped anastomosis
Procedure: Handsewn anastomosis — a handsewn anastomosis technique will be used during fistula creation.
  Arms: Handsewn anastomosis

SUMMARY:
The purpose of this study is to determine whether handsewn anastomosis versus clipped technique is associated with more complications, fistula failures, surgical cost and surgical time.

DETAILED DESCRIPTION:
End stage renal disease requiring hemodialysis has become more prevalent in recent years. Achieving vascular access is an important step in receiving hemodialysis. Recent national goals have established that approximately 65% of all dialysis access points should be arteriovenous fistulas due to higher patency rates and decreased rates of further surgeries. Multiple studies have been done to assess optimal suture technique for arteriovenous anastomoses. The use of clips versus a handsewn technique has been evaluated in retrospective studies with some reports indicating a higher primary patency rate with a clip technique. Further study is needed to definitively determine the technique that results in the highest patency rates and lowest rate of re-operation. The purpose of this study is to determine whether hand-sewn anastomosis versus a clipped technique is associated with more complications, failures, surgical cost and surgical time by randomizing patients to either a clipped anastomosis group or a handsewn anastomosis group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Need for AVF creation for vascular access for planned hemodialysis (within 1 year).
* The planned AVF site must be naïve of prior AVF creations.
* Vein mapping studies completed
* 2.5 - 3mm minimum vein diameter on mapping

Exclusion Criteria:

* Less than 18 years of age.
* Inability to provide consent.
* Previous failed AVFs in both arms.
* Contraindications to AVF creation:

  * ipsilateral proximal venous and arterial occlusion or stenosis
  * systemic or local infection
  * too ill to operate
* Anticipated inability to keep 30-day postoperative follow-up appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patency rates | 2 years postoperative
  Patency will be assessed and the fistula considered patent if it has been accessed for dialysis at least once, or based on clinical assessment with palpable thrill if dialysis access has not been attempted.

SECONDARY OUTCOMES:
Surgical complications | 2 years postoperative
  Complications will be monitored intraoperatively, and postoperatively. These include any re-interventions, and wound complications, infection, hematoma, thrombosis , steal syndrome, distal ischemia.

OTHER OUTCOMES:
Cost | 1 year postoperative
  Cost for the vascular clip device will be compared to cost of the handsewn technique.

CONTACTS AND LOCATIONS:
Overall Officials: Clark A Davis, MD, Principal Investigator — Gundersen Lutheran Health System
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States

REFERENCES:
- [Background] Baguneid MS, Goldner S, Fulford PE, Hamilton G, Walker MG, Seifalian AM. A comparison of para-anastomotic compliance profiles after vascular anastomosis: nonpenetrating clips versus standard sutures. J Vasc Surg. 2001 Apr;33(4):812-20. doi: 10.1067/mva.2001.112806. PMID 11296337
- [Background] Lin PH, Bush RL, Nelson JC, Lam R, Paladugu R, Chen C, Quinn G, Lumsden AB. A prospective evaluation of interrupted nitinol surgical clips in arteriovenous fistula for hemodialysis. Am J Surg. 2003 Dec;186(6):625-30. doi: 10.1016/j.amjsurg.2003.08.007. PMID 14672769
- [Background] Varcoe RL, Teo AB, Pelletier MH, Yu Y, Yang JL, Crowe PJ, Walsh WR. An arteriovenous fistula model of intimal hyperplasia for evaluation of a nitinol U-Clip anastomosis. Eur J Vasc Endovasc Surg. 2012 Feb;43(2):224-31. doi: 10.1016/j.ejvs.2011.11.002. Epub 2011 Nov 21. PMID 22104322
- [Background] Shenoy S, Miller A, Petersen F, Kirsch WM, Konkin T, Kim P, Dickson C, Schild AF, Stewart L, Reyes M, Anton L, Woodward RS. A multicenter study of permanent hemodialysis access patency: beneficial effect of clipped vascular anastomotic technique. J Vasc Surg. 2003 Aug;38(2):229-35. doi: 10.1016/s0741-5214(03)00412-9. PMID 12891102
- [Background] Shenoy S, Woodward RS. Economic impact of the beneficial effect of changing vascular anastomotic technique in hemodialysis access. Vasc Endovascular Surg. 2005 Sep-Oct;39(5):437-43. doi: 10.1177/153857440503900509. PMID 16193217